CLINICAL TRIAL: NCT04395911
Title: A Multi-Center Pilot Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device (SCD) in Patients Developing Acute Kidney Injury (AKI) or Acute Respiratory Distress Syndrome (ARDS) Associated With COVID-19 Infection
Brief Title: Safety and Efficacy of SCD in AKI or ARDS Patients Associated With COVID-19 Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SeaStar Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCD-005
Record Dates: First submitted 2020-05-17; First posted 2020-05-20 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: AKI; ARDS; COVID

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SCD (Other): Cytopheretic device
  Interventions: Device: SCD

INTERVENTIONS:
Device: SCD — cytopheretic device

SUMMARY:
Selective Cytopheretic Device (SCD) treatments will improve survival in patients testing positive for COVID-19 infection diagnosed with Acute Kidney Injury (AKI) or ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Positive COVID-19 test
* Must be receiving medical care in an intensive care nursing situation
* Non-pregnant females
* Intent to deliver full supportive care through aggressive management utilizing all available therapies for a minimum of 96 hours.
* Platelet count >30,000/mm3 at Screening
* Clinical diagnosis of AKI requiring CRRT or ARDS

Exclusion Criteria:

* Cardiovascular instability that precludes initiation of continuous renal replacement therapy (CRRT).
* Irreversible brain damage based on available historical and clinical information.
* Presence of any solid organ transplant at any time.
* Patients with stem cell transplant in the previous 100 days or who have not engrafted.
* Acute or chronic use of circulatory support device other than ECMO such as LVADs, RVADs, BIVADs.
* Metastatic malignancy which is actively being treated or may be treated with chemotherapy or radiation during the subsequent three month period after study treatment.
* Chronic immunosuppression defined as >20 mg prednisone qd alone without other immunosuppressant medications (ie (cyclophosphamide, azathioprine, methotrexate, rituximab, mycophenolate, cyclosporine).
* Patient is moribund or chronically debilitated for whom full supportive care is not indicated.
* Concurrent enrollment in another interventional clinical trial. Patients enrolled in observational studies (NO TEST DEVICE OR DRUG USED) are allowed to participate.
* Any reason the Investigator deems exclusionary.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Mortality at Day 60 | 60 days post treatment
  All cause mortality at Day 60
Dialysis Dependency | 60 days post treatment
  Dialysis Dependency at Day 60
Ventilation at Day 28 | 28 days post treatment
  Ventilation free survival at Day 28

SECONDARY OUTCOMES:
Dialysis Dependency | 28 days post treatment
  Dialysis Dependency at Day 28
Mortality at Day 28 | 28 days post treatment
  All cause mortality at Day 28
Urinary output change | 10 days of treatment
  Change from baseline in urine output
P02/FiO2 change | 10 days of treatment
  Change from baseline in PO2/FiO2
Safety Assessments | 10 days of treatment
  Assessment of SAEs, AE and UADEs
SCD Integrity | 10 days of treatment
  Assessment of device performance

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Unidentified participant data collected for this study will be submitted to a CRO for data analysis. All data will be submitted to the Sponsor.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be collected throughout the study conduct.
Access Criteria: Participant data will be accessible to the Investigational Site and CRO through a secured electronic data capture system. CRO personnel will be responsible for data verification. De-identified Participant information will be accessible to the CRO and the Sponsor.